CLINICAL TRIAL: NCT01212939
Title: Revitalization of Teeth With Necrotic Pulps and Open Apexes Using Platelet-Rich Plasma
Status: Terminated | Type: Observational
Why Stopped: No advantage seen during continued animal studies. Difficult recruitment.
Sponsor: Torabinejad, Mahmoud (Other)
Responsible Party: Sponsor-Investigator, Torabinejad, Mahmoud, Principal Investigator, Loma Linda University
Organization: Loma Linda University (Other)
Other Study IDs: IRB# 5100239
Record Dates: First submitted 2010-09-29; First posted 2010-10-01 (Estimated); Last update posted 2014-04-04 (Estimated); Status verified 2014-04

CONDITIONS: Infection
Keywords: Dead pulps and open root ends; Patients who have teeth with dead pulp and open root ends
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
When root canals of infected teeth with closed ends are cleaned, disinfected and filled, the results are predictable with excellent outcomes. However, in a tooth with incomplete root development, the end of the root(s) must be closed before filling the root canals. One or two-step artificial barrier using mineral trioxide aggregate (MTA) has been used before filling the root canals of these teeth. Despite the high success of this treatment, this procedure does not result in complete root formation and these teeth are susceptible to root fracture. A number of case reports in scientific journal have shown the possibility for regeneration of nerve within the root canal space and continued root development in teeth with dead nerves and open ends. There is very little information regarding the use of stem cells and growth factors from the blood of patients to regenerate the nerves in these teeth. Platelet rich plasma (PRP) from whole blood has been mentioned in the literature as a potential ideal material for regeneration of nerves in these teeth. The purpose of this study is to investigate the use of PRP to regenerate tooth nerve and close the root ends in teeth with root canal infection and open root ends.

DETAILED DESCRIPTION:
Procedures Participants in this study must be in overall good health and not allergic to the materials used during this study treatment. If you agree to participate in this study, you will receive a screening visit to determine whether you will qualify for the study. At that time, your medical history will be reviewed, your blood pressure and pulse will be taken and you will be asked to fill out detailed medical and dental histories. In addition, you will receive an examination of your teeth and gums.

In the first appointment, after anesthetizing you with a local anesthetic similar to Novocain and application of a rubber dam to isolate your tooth, an opening will be made into the root canal(s). The canal(s) will be cleaned and medicated with antibiotics to get rid of the infection and sealed with a temporary filling material. Except for the use of antibiotics the rest of the procedures done in this appointment are similar to what the investigators do for the patients for need root canal treatment.

In the second appointment, after providing anesthesia with Novocain and application of rubber dam again, the temporary filling will be removed and the antibiotic will be removed using sterile water. The canal will be then dried. During this appointment, 20 ml of whole blood will be taken from your arm vein and will be used to prepare concentrated cells for injection into the prepared canal and sealed again with a temporary filling material. This part is different than what the investigators normally do for patients who need root canal treatment. For those patients the investigators fill the canals and seal the opening into the root canals with a permanent filling material.

You will return three to seven days later to the endodontic clinic and at that time, after rubber dam application, the temporary filling material will be removed and the tooth will be double sealed with permanent filling materials. This is an extra step that the investigators normally do not take for patients who need root canal treatment. A dental assistant or a dentist will call you to make an appointment at 3, 6, 12, 18, and 24 months following completion of your root canal treatment to check the vitality of the tooth using an ice stick and closure of the root end. Checking the process of healing in your tooth is similar to what the investigators routinely do for our patients who require root canal treatment.

Risks The study will require drawing blood from your arm. Veins and arteries vary in size from one person to another and from one side of the body to the other. Obtaining a blood sample from some people may be more difficult than from others. Other risks associated with having blood drawn are slight but may include bleeding, fainting or feeling light-headed, hematoma (blood accumulating under the skin), and infection (a slight risk any time the skin is broken). In rare instances, it may cause severe pain of infection. Depending upon the complications, your dentist may decide to remove the PRP completely out of the root canal and the use other procedures to treat your tooth. Should root canal failure occur, further dental treatment will be rendered at no charge to you.

Benefits Whether or not you will benefit from this study is not yet known. However, there is a possibility of saving the tooth with this procedure. Your participation will help dentists learn about the importance of regeneration of nerves in teeth with infection and open root ends, and may help save your tooth.

Participants' Rights Your participation in this study is voluntary. Your decision whether or not to participate or terminate at any time will not affect your present or future treatment here at the Dental School. You may withdraw from the study at any time that you want to.

Alternative Treatments You can choose not to participate in this study and have your tooth treated with the standard root canal procedures or have it extracted. Refusal to participate in this study will involve no penalties or loss of usual benefits to which you are entitled.

Confidentiality The medical information collected in this study will be available to the investigators, the U.S. Food and Drug Administration, and the Institutional Review Board of Loma Linda University. The results may be published but your name will not be used in publications. However, submission of the information will be accomplished with strict adherence to the professional standards of confidentiality. See attached PHI Authorization for more information about your privacy. Your name and address will be kept on record at the investigator's office in case you need to be contacted in the future about this study.

ELIGIBILITY:
Inclusion Criteria:

* People with necrotic pulp and open apex.

Exclusion Criteria:

* People with vital pulp and closed apexes

Ages: 6 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients between the ages of 6-89
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2012-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
stop the infection | 6 weeks

SECONDARY OUTCOMES:
Revitalizing the nerve of the tooth | Every 3-6 months for two years

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Torabinejad, DDS, Principal Investigator — Loma Linda University
Locations (2):
- United States (2):
  - Loma Linda Dental School, Loma Linda, California
  - Loma Linda University, Loma Linda, California